CLINICAL TRIAL: NCT04008771
Title: A Phase 1 Safety And Effectiveness Study of Intravitreal Injection of SeeQ CdSe 655 Alt Nanoparticles for Patients With Degenerative Retinal Diseases
Brief Title: Intravitreal Injection of SeeQ CdSe 655 Alt Nanoparticles for Patients With Degenerative Retinal Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 2C Tech Corp (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SeeQ 101.A
Record Dates: First submitted 2019-06-25; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: This study was a prospective, open label feasibility study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Severe Disease (Experimental): Subjects with baseline BCVA between 20/16000 and hand motion (HM). Subjects received 2.0 μM concentration intravitreal injections on each Day 0 and Day 21.
  Interventions: Device: SeeQ CdSe 655 ALT
- Moderate to Severe Disease (Experimental): Subjects with baseline BCVA from 20/60 to 20/16000. The first five (5) to receive 2.0 μM concentration intravitreal at each Day 0 and Day 21, the subsequent five (5) to receive 0.2 μM intravitreal injection at each Day 0 and Day 21, additional subjects (up to ten [10]) to receive one of the dosing options (either 2.0 μM or 0.2 μM) at each Day 0 and Day 21, at the discretion of the Investigator and Sponsor.
  Interventions: Device: SeeQ CdSe 655 ALT

INTERVENTIONS:
Device: SeeQ CdSe 655 ALT — SeeQ CdSe 655 Alt is a sterile colloidal solution of coated CdSe nanoparticles in a borate buffer suitable for intraocular injection.

SUMMARY:
This study was a prospective, open label feasibility study conducted at a single clinical site (APEC, Mexico City) to evaluate the safety and preliminary effectiveness of the SeeQ device, with each patient's serving as his/her own contralateral control.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 21 years of age or older.
2. Subjects with a history of degenerative retinal diseases such as RP.
3. Subjects with a documented history of disease progression.
4. Willing and able to return for all study visits.
5. Willing and able to provide written informed consent for the Clinical Study.
6. Subjects with a BCVA greater or equal to 20/16000 must have consistent fixation demonstrated by indirect ophthalmoscopy with a small circle of light and by consistent location of remaining central visual field detected by VFA.
7. Study Arm A: The best corrected visual acuity must be between 20/16000 and HM as tested by ETDRS chart and ERG B wave amplitude.
8. Study Arm B: The best-corrected visual acuity must be between 20/60 and 20/16000 and visual field of central 15 degrees (III static 30-2 protocol, 31.5 ASB background) greater than 10 dB loss, as determined by a Humphrey Instruments, Inc. Visual Field Analyzer (VFA).

Exclusion Criteria:

1. Subjects with significant lens or corneal pathology (either history of or current) in the study eye other than retinal diseases.
2. Subjects with high myopia in the study eye (axial length greater than or equal to 26.0 millimeters by ultrasound or spherical equivalent at the spectacle plane greater than -8.0 diopters.)
3. Subjects whose retinal disease status has been stable for more than 90 days.
4. Subjects with history of iritis or uveitis in either eye.
5. Subjects who have monocular vision.
6. Subjects with a history of retinal detachment or tear in either eye.
7. Subjets with unstable IOP (i.e. > 30 mmHg in the past six months) or IOP of > 24 mm Hg at enrollment while under medical control. Subjects may be on topical medications to control their IOP.
8. Subjects with an aphakic study ete or if pseudophakic, cataract extraction surgery more than 6 months prior to study enrollment.
9. Subjects with a history of ocular trauma of any type in the study eye.
10. Subjects with media opacities or abnormalities that would preclude observation of the retina in the study eye, per the investigator's judgement.
11. Subjects that have undergone any previous vitrectomy (either anterior or pars plana vitrectomy in the study eye).
12. Subjects with a history of cataract surgery complication in the study eye.
13. Subjects that have undergone previous photocoagulation of the retina in the study eye.
14. Subjects anticipated requiring cataract extraction in the study eye within the next six (6) months.
15. Subjects with congenital eye malformations.
16. Recurrent uveitis or history of uveitis in either eye.
17. Macular edema or history of macular edema in the study eye where central macular thickness is greater than 275 microns by OCT at baseline.
18. Ongoing ocular infection or inflammation in the study eye.
19. Pregnant or nursing females.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2014-12-19 (Actual); Study Completion 2014-12-19 (Actual)

PRIMARY OUTCOMES:
Change in Best Corrected Visual Acuity "BCVA" | Measured at Baseline through Day 42
Change in Contrast Sensitivity | Measured at Baseline through Day 42
  Contrast sensitivity was measured utilizing a sin wave (Vistech) contrast sensitivity chart under photopic conditions
Change in ERG Amplitude | Measured at Baseline through Day 42
  ERG amplitude was measured using Poland Consult ERG equipment
Change in Visual Fields | Measured at Baseline through Day 42
  Visual Field improvement is assessed using a Humphrey/Zeiss Visual Field Analyzer
Change in Functional Vision | Measured at Baseline through Day 42
  Functional Vision is tested using Object identification and White line orientation testing

SECONDARY OUTCOMES:
Duration of Effect | Measured at Baseline through Day 42

OTHER OUTCOMES:
Rate of Ocular Adverse Events | Measured at Baseline through Day 42
  Safety Endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Asociacion Para Evitar La Ceguera En Mexico, I.A.P. (APEC), Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No